CLINICAL TRIAL: NCT04116619
Title: Investigating Stress-related Mechanisms in the Laboratory and Real World in Individuals With Cannabis Use Disorder
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Stephanie Wemm, Associate Research Scientist, Yale University
Other Study IDs: 2000026364; KL2TR001862 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Cannabis Use Disorder: Participants who meet criteria for Cannabis Use Disorder will complete three guided imagery conditions (stress, cannabis, neutral) in an inpatient research unit. During the guided imagery, repeated measurements of subjective (i.e., craving, negative affect), neuroendocrine (i.e., cortisol), and physiological variables (i.e., heart rate variability [HRV]) will be collected.
  Interventions: Other: Guided Imagery Laboratory Session
- Light Cannabis Users: Participants who are light cannabis users (<1 joint/week) will complete three guided imagery conditions (stress, cannabis, neutral) in an inpatient research unit. During the guided imagery, repeated measurements of subjective (i.e., craving, negative affect), neuroendocrine (i.e., cortisol), and physiological variables (i.e., heart rate variability [HRV]) will be collected.
  Interventions: Other: Guided Imagery Laboratory Session

INTERVENTIONS:
Other: Guided Imagery Laboratory Session — On days 1, 2 and 3 of the study, subjects will come to the research testing rooms and be provided with lunch before beginning the laboratory session. After a 40-minute adaptation period, two blood samples will be drawn before imagery (BASELINE). After the second blood draw, a 5-minute baseline period will follow to assess continuous pulse rate, BP, and HRV assessments. The subject and research staff conducting the sessions will be blinded to the order and content of the imagery condition. In each recording, the subjects will listen to the scripts over headphones and will vividly imagine the described situation, 'as if' it were happening right now," for 5 minutes. The research nurse will take a blood draw immediately after the imagery (IMAGERY). After that, three recovery blood draws will be performed at 15-minute intervals (RECOVERY). We will analyze the total of six blood samples for levels of cortisol.

SUMMARY:
This research project proposes a novel approach to elucidate the biological adaptations associated with Cannabis Use Disorder and to assess whether such adaptations are predictive of higher drug craving in response to both drug cues and stressors in both the laboratory and real-world, and higher relapse risk and drug use in the real world.

DETAILED DESCRIPTION:
The intent of this study is to recruit 25 treatment-seeking individuals with Cannabis Use Disorder (CUD) and 25 light users (<1 joint/week) to complete three guided imagery conditions (stress, cannabis, neutral) in inpatient research units. During the guided imagery, repeated measurements of subjective (i.e., craving, negative affect), neuroendocrine (i.e., cortisol), and physiological variables (i.e., heart rate variability [HRV]) will be collected. Thereafter, individuals with CUD will begin one-month of drug counseling treatment coupled with surveys delivered via smartphones daily in the morning, evening, and at four random times during the day.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis using men and women who:
* 1. Are fluent in English;
* 2. Are using cannabis at levels to match either of the two groups:

  a) Light Users: i. Cannabis using levels of < 1 joint/week ii. Has never met DSM-5 criteria for CUD or other substance use disorders. b) Individuals with Cannabis Use Disorder: i. Meets criteria for CUD based on the SCID (≤ 2 symptoms in past year); ii. Has a past-year cannabis use pattern of ≤3 times per week; iii.Do not meet criteria for any other substance use disorders other than mild Alcohol Use Disorder.
* 3. Provide a negative breathalyzer for alcohol and only positive for cannabis use at all appointments;
* 4. Can provide written informed consent.

Exclusion Criteria:

* 1. Meets current or past DSM-5 criteria for Axis I for major psychiatric disorders, other than depression or anxiety disorder;
* 2. Meets criteria for a current Substance Use Disorder other than Cannabis or mild Alcohol Use Disorder;
* 3. Has any significant current medical conditions requiring medication, including neurological, renal, thyroid, cardiovascular, liver, endocrine, or immune conditions;
* 4. Reports current use of medications/drugs that interfere with HPA axis response,
* 5. Are women who are pregnant or lactating, are peri-/post-menopausal, or those with hysterectomies;
* 6. Report current use of psychotropic drugs other than antidepressants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with Cannabis Use Disorder and individuals who use cannabis <1/week and do not meet criteria for Cannabis Use Disorder
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Rating of craving in the laboratory | 3 days
  Participants will rate their level of stress and marijuana craving at five time points during the laboratory session, once at pre-baseline, baseline, immediately post-imagery procedures, and at three times point 15, 30, and 45 minutes post-imagery. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High." Individuals with CUD will be compared to light marijuana users in their differences in slope in response to the imagery.
Rating of subjective stress in the laboratory | 3 days
  Participants will rate their level of stress and marijuana craving at five time points during the laboratory session, once at pre-baseline, baseline, immediately post-imagery procedures, and at three times point 15, 30, and 45 minutes post-imagery. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High." Individuals with CUD will be compared to light marijuana users in their differences in slope in response to the imagery.
Rating of subjective craving in the real world | 28 days
  Participants will report using ecological momentary assessment (EMA) their current levels of stress and craving, if they have used marijuana, and if they experienced a stressor. These reports will be generated in three different ways: at 8 am and 8 pm at night, at four random times during waking hours, and during marijuana use. Individuals with CUD will be compared to light marijuana users in their differences in real-world ratings of stress and craving. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High."
Rating of subjective stress in the real world | 28 days
  Participants will report using ecological momentary assessment (EMA) their current levels of stress and craving, if they have used marijuana, and if they experienced a stressor. These reports will be generated in three different ways: at 8 am and 8 pm at night, at four random times during waking hours, and during marijuana use. Individuals with CUD will be compared to light marijuana users in their differences in real-world ratings of stress and craving. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High."
Physiological response to stress and cannabis cues in the laboratory | 3 days
  Plasma will be collected at each laboratory session to assess cortisol response to stress, drug cue, and neutral imagery exposure. Heart Rate Variability (HRV) measured via the Firstbeat Bodyguard 2 will be used to assess cardiovascular response to stress, drug, and neutral cue imagery exposure.
Heart rate response to stress and cannabis cues in the real world | 2 weeks
  Heart Rate Variability (HRV) will be collected throughout the day on two separate three-day occasions during Weeks 1 and Week 2 via the Firstbeat Bodyguard.

SECONDARY OUTCOMES:
Blood pressure- diastolic | 2 weeks
  A General Electric Dynamap will be used to place a blood pressure cuff on the subject's preferred arm to monitor blood pressure (BP) during the laboratory sessions in week 2 in order to assess change in BP responses to stress, drug cue and neutral provocation.
Blood pressure- systolic | 2 weeks
  A General Electric Dynamap will be used to place a blood pressure cuff on the subject's preferred arm to monitor blood pressure (BP) during the laboratory sessions in week 2 in order to assess change in BP responses to stress, drug cue and neutral provocation.
Change in Cannabis use- Labs | 4 weeks
  Cannabis use will be determined using a urine toxicology screen. Change in percent THCCOOH levels assessed via urine during the 4 week trial assessed by a weekly urine toxicology screen.
Change in Cannabis use- Self Report | 4 weeks
  Change over time in daily reporting of cannabis use per day will be assessed by self-report on the Timeline Followback.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wemm, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No